CLINICAL TRIAL: NCT00293397
Title: Treatment of Patients With Hepatocellular Carcinoma Using Drug-Eluting Bead Embolization
Brief Title: Chemoembolization Using Doxorubicin in Treating Patients With Liver Cancer That Cannot Be Removed By Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000456493; P30CA006973 (NIH); JHOC-J0516; HOC-05042805
Record Dates: First submitted 2006-02-16; First posted 2006-02-17 (Estimated); Results first posted 2018-07-18 (Actual); Last update posted 2018-07-18 (Actual); Status verified 2018-06

CONDITIONS: Liver Cancer
Keywords: adult primary hepatocellular carcinoma; localized unresectable adult primary liver cancer
MeSH Terms: conditions — Liver Neoplasms; Carcinoma, Hepatocellular

ARMS (1):
- Drug-eluting bead transarterial chemoembolization (DEB-TACE) (Experimental): Patients undergo DEB-TACE procedures utilizing LC Beads, polyvinyl alcohol microspheres with diameters of 100-300um or 300-500um, which are loaded with 100mg of doxorubicin hydrochloride and mixed with an equal volume of nonionic contrast media.
  Interventions: Device: Drug-eluting beads loaded with doxorubicin hydrochloride

INTERVENTIONS:
Device: Drug-eluting beads loaded with doxorubicin hydrochloride — Doxorubicin eluting beads
  Other Names: Gelspheres; LC Beads

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as doxorubicin, work in different ways to stop the growth of tumor cells, either by killing the cells or stopping them from dividing. Chemoembolization kills tumor cells by blocking the blood flow to the tumor and keeping chemotherapy drugs near the tumor.

PURPOSE: This clinical trial is studying how well chemoembolization using doxorubicin works in treating patients with liver cancer that cannot be removed by surgery.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine, preliminarily, the feasibility of chemoembolization with GelSpheres™ beads mixed with doxorubicin hydrochloride in patients with unresectable hepatocellular carcinoma.

OUTLINE: This is a pilot study.

Patients undergo catheterization of the hepatic artery followed by chemoembolization comprising an infusion of GelSpheres™ beads mixed with doxorubicin hydrochloride into the target hepatic artery. Patients may receive up to 3 chemoembolization treatments.

After completion of study treatment, patients are followed at 1 month, every 2 months for 1 year, and then every 3 months during year 2.

PROJECTED ACCRUAL: A total of 20 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of hepatocellular carcinoma (HCC) according to the European Association for the Study of Liver (EASL) disease diagnostic criteria AND the Okuda staging classification

  * No advanced disease, as defined by any of the following:

    * Barcelona Clinic Liver Cancer (BCLC) class C disease, as defined by the following:

      * Vascular invasion, including segmental portal obstruction
      * Extrahepatic spread
      * Cancer-related symptoms (PST of 1-2)
    * BCLC class D disease, as defined by the following:

      * Okuda stage III disease
      * World Health Organization (WHO) performance status 3 or 4
    * Diffuse HCC, defined as massive ill-defined tumor involvement
    * Child-Pugh Class C
* Not eligible for radical therapies (e.g., resection, liver transplantation, or percutaneous therapies)
* No significant liver decompensation

  * Preserved liver function (Child-Pugh class A-B)

    * No ascites (trace ascites allowed)
* No other active primary tumor
* Arteries supplying the lesion must be large enough to accept GelSpheres™ beads

PATIENT CHARACTERISTICS:

* Bilirubin ≤ 3 mg/dL
* Albumin > 2.0 g/dL
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 5 times the upper limit of normal (ULN)
* Alkaline phosphatase ≤ 5 times the upper limit of normal (ULN)
* No active gastrointestinal bleeding
* No encephalopathy
* No contraindication to hepatic embolization procedures, as indicated by any of the following:

  * Porto-systemic shunt
  * Hepatofugal blood flow
  * Platelet count < 50,000/mm^3
  * International normalized ratio (INR) ≥ 1.8
  * Partial thromboplastin time (PTT) ≥ 39 seconds
  * Renal failure
  * Severe atheromatosis
* No contraindication to doxorubicin hydrochloride administration, as indicated by any of the following:

  * Bilirubin > 5 mg/dL
  * White blood cell (WBC) < 1,500/mm^3
  * Ejection fraction < 50% by isotopic ventriculography or echocardiography
* Not pregnant
* No known allergy to contrast media
* No intolerance to occlusion procedures
* No vascular anatomy or bleeding that would preclude catheter placement or emboli injection, as indicated by any of the following:

  * Active or risk of hemorrhage
  * Patent extra-to-intracranial anastomoses or shunts
  * End arteries leading directly to the cranial nerves
  * Feeding arteries smaller than distal branches from which they emerge
  * Collateral vessel pathways that would potentially endanger normal territories during embolization

PRIOR CONCURRENT THERAPY:

* No prior anticancer therapy for HCC

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2005-11; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey F. Geschwind, MD, Study Chair — Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins
Locations (1):
- Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland, United States

REFERENCES:
- [Result] Reyes DK, Vossen JA, Kamel IR, Azad NS, Wahlin TA, Torbenson MS, Choti MA, Geschwind JF. Single-center phase II trial of transarterial chemoembolization with drug-eluting beads for patients with unresectable hepatocellular carcinoma: initial experience in the United States. Cancer J. 2009 Nov-Dec;15(6):526-32. doi: 10.1097/PPO.0b013e3181c5214b. PMID 20010173

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 20 patients with unresectable hepatocellular carcinoma (HCC) were enrolled at Johns Hopkins Hospital to undergo treatment with drug-eluting beads (DEBs) infused with doxorubicin. The last patient was enrolled in Dec 2007.
Groups:
- Drug-eluting Bead Transarterial Chemoembolziation (DEB-TACE): Patients undergo DEB-TACE procedures utilizing LC Beads, polyvinyl alcohol microspheres with diameters of 100-300um or 300-500um, which are loaded with 100mg of doxorubicin hydrochloride and mixed with an equal volume of nonionic contrast media.
  doxorubicin hydrochloride: Doxorubicin eluting beads
Period: Overall Study
Arm/Group | Drug-eluting Bead Transarterial Chemoembolziation (DEB-TACE)
Started | 20
Received First DEB-TACE | 19 (1 patient death after baseline inclusion screening and before first treatment)
Completed | 18 (1 patient death within 30 days post-TACE - not attributed to TACE procedure)
Not Completed | 2
Not completed — Death | 2

BASELINE CHARACTERISTICS:
Arm/Group | Drug-eluting Bead Transarterial Chemoembolziation (DEB-TACE)
Number analyzed (Participants) | 20
Age, Continuous [Mean (Full Range); unit: years] | 64 [41 to 85]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 12
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 20
Barcelona Clinic Liver Cancer (BCLC) grade [Count of Participants; unit: Participants] — The Barcelona Clinic Liver Cancer (BCLC) grades are used to assess those with Hepatocellular carcinoma (HCC). Grade A is the least severe, grade B is moderate and grade C is advanced.
  Participants
    BCLC A | 6
    BCLC B | 2
    BCLC C | 12

OUTCOME MEASURES:

1. Primary Outcome: Safety
Description: Safety was assessed using the CTCAE v 3.0 criteria, reported are the number of participants that experienced at least 1 event that was grade 2 (moderate) or higher.
Time Frame: 1 month
Population: 19 of 20 patients were assessed at 1 month.
Measure: Count of Participants; unit: Participants
Arm/Group | Drug-eluting Bead Transarterial Chemoembolziation (DEB-TACE)
Number analyzed (Participants) | 19
Participants
  Grade 2 | 16
  Grade 3 | 3

2. Primary Outcome: Safety
Description: as for outcome 1
Time Frame: 6 months
Population: 19 of 20 patients were assessed at 6 months.
Measure: Count of Participants; unit: Participants
Arm/Group | Drug-eluting Bead Transarterial Chemoembolziation (DEB-TACE)
Number analyzed (Participants) | 19
Participants
  Grade 2 | 8
  Grade 3 | 1

3. Primary Outcome: Efficacy - Tumor Response by the European Association for the Study of the Liver (EASL) Criteria
Description: Efficacy as assessed by radiographic tumor response using EASL criteria at baseline and at 1 month post-TACE
  Complete Response (CR): Achieving 100% tumor necrosis of targeted lesions Partial Response (PR): Demonstrating greater than 50% tumor necrosis in targeted lesions Progressive Disease (PD): Reappearance of or increased tumor enhancement greater than 25% in targeted lesions Stable Disease (SD): Not meeting requirements for CR or PR and not demonstrating evidence of progression in targeted lesions.
Time Frame: 1 month
Population: 19 of 20 patients were assessed at 1 month.
Measure: Count of Participants; unit: Participants
Groups:
- Drug-eluting Bead Transarterial Chemoembolization (DEB-TACE): Patients undergo DEB-TACE procedures utilizing LC Beads, polyvinyl alcohol microspheres with diameters of 100-300um or 300-500um, which are loaded with 100mg of doxorubicin hydrochloride and mixed with an equal volume of nonionic contrast media.
  doxorubicin hydrochloride: Doxorubicin eluting beads
Arm/Group | Drug-eluting Bead Transarterial Chemoembolization (DEB-TACE)
Number analyzed (Participants) | 19
Participants
  1 month post-TACE : Complete Response (CR) | 6
  1 month post-TACE : Partial Response (PR) | 6
  1 month post-TACE : Stable Disease (SD) | 8
  1 month post-TACE : Progressive Disease | 0
  Disease control rate (CR + PR + SD) | 19

4. Primary Outcome: Efficacy - Tumor Response by Response Evaluation Criteria in Solid Tumors (RECIST)
Description: Efficacy as assessed by radiographic tumor response using RECIST criteria at baseline, 1 month post treatment.
  Complete Response (CR): Disappearance of all lesions targeted by therapy Partial Response (PR): At least 30% decrease in the sum of longest diameter (LD) of lesions targeted by therapy Progressive Disease (PD): At least 20% increase in sum of LD of lesions targeted by therapy Stable Disease (SD): Neither sufficient shrinkage for PR nor sufficient increase for PD.
Time Frame: 1 month
Population: 19 of 20 patients were assessed at 1 month.
Measure: Count of Participants; unit: Participants
Arm/Group | Drug-eluting Bead Transarterial Chemoembolization (DEB-TACE)
Number analyzed (Participants) | 19
Participants
  1 month post-TACE : Complete Response (CR) | 0
  1 month post-TACE : Partial Response (PR) | 2
  1 month post-TACE : Stable Disease (SD) | 18
  1 month post-TACE : Progressive Disease | 0
  Disease control rate (CR + PR + SD) | 19

5. Primary Outcome: Efficacy - Tumor Response by Response Evaluation Criteria in Solid Tumors (RECIST)
Description: Efficacy as assessed by radiographic tumor response using RECIST criteria at baseline, and at 6 months post treatment.
  Complete Response (CR): Disappearance of all lesions targeted by therapy Partial Response (PR): At least 30% decrease in the sum of longest diameter (LD) of lesions targeted by therapy Progressive Disease (PD): At least 20% increase in sum of LD of lesions targeted by therapy Stable Disease (SD): Neither sufficient shrinkage for PR nor sufficient increase for PD.
Time Frame: 6 months
Population: 19 of 20 patients were assessed.
Measure: Count of Participants; unit: Participants
Arm/Group | Drug-eluting Bead Transarterial Chemoembolization (DEB-TACE)
Number analyzed (Participants) | 19
Participants
  6 months post-TACE : Complete Response (CR) | 1
  6 months post-TACE : Partial Response (PR) | 7
  6 months post-TACE : Stable Disease (SD) | 11
  6 months post-TACE : Progressive Disease (PD) | 1
  Disease control rate (CR + PR + SD) | 19

6. Primary Outcome: Efficacy - Overall Survival
Description: Presented are the counts of patients that have survived up to 1 year.
Time Frame: 1 Year
Population: 20 patients were assessed.
Measure: Count of Participants; unit: Participants
Arm/Group | Drug-eluting Bead Transarterial Chemoembolization (DEB-TACE)
Number analyzed (Participants) | 20
Participants | 13

7. Primary Outcome: Efficacy - Overall Survival
Description: Presented are the counts of patients that have survived up to 2 years.
Time Frame: 2 Years
Population: 20 patients were assessed.
Measure: Count of Participants; unit: Participants
Arm/Group | Drug-eluting Bead Transarterial Chemoembolization (DEB-TACE)
Number analyzed (Participants) | 20
Participants | 11

ADVERSE EVENTS:
Time Frame: 3 months
Arm/Group | Drug-eluting Bead Transarterial Chemoembolziation (DEB-TACE)
All-Cause Mortality (participants affected / at risk) | 2/20
Serious Adverse Events (participants affected / at risk) | 2/20
Other Adverse Events (participants affected / at risk) | 20/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Drug-eluting Bead Transarterial Chemoembolziation (DEB-TACE) (N=20)
Liver failure (Hepatobiliary disorders) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Drug-eluting Bead Transarterial Chemoembolziation (DEB-TACE) (N=20)
Fatigue (General disorders) | 13 (13)
Post-embolization syndrome (Gastrointestinal disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 8 (8)
Fever (General disorders) | 3 (3)
Nausea (Gastrointestinal disorders) | 3 (3)
Vomiting (Gastrointestinal disorders) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 9 (9)
Leukocytopenia (Investigations) | 5 (5)
Thrombocytopenia (Investigations) | 3 (3)
Elevated liver enzymes (Investigations) | 6 (6)
Anorexia (Metabolism and nutrition disorders) | 7 (7)
Weight loss (Investigations) | 6 (6)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1)
Decreased libido (Psychiatric disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Gastroenteritis (Gastrointestinal disorders) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes